CLINICAL TRIAL: NCT01803503
Title: Phase II Randomized Study of Docetaxel With or Without Low-dose, Short Course Sunitinib in the Treatment of Advanced Solid Tumors
Brief Title: Docetaxel With or Without Low-dose, Short Course Sunitinib in Refractory Solid Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BR01/08/13; 2013/00170 (Other: NHG Domain Specific Review Boards)
Record Dates: First submitted 2013-03-01; First posted 2013-03-04 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Solid Tumors; Breast Cancer; Non-small Cell Lung Cancer; Prostate Cancer; Gastric Cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Prostatic Neoplasms; Stomach Neoplasms | interventions — Docetaxel; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Docetaxel (Active Comparator): Docetaxel 75mg/m2 day 1, every 3 weeks. Patients will be treated for a maximum of 6 cycles of chemotherapy in the absence of tumor progression or unacceptable toxicities.
  Interventions: Drug: Docetaxel
- Docetaxel + Sunitinib (Experimental): Docetaxel 75mg/m2 day 1, every 3 weeks, preceded by 7 days of sunitinib 12.5mg orally daily during each cycle.
  Patients will be treated for a maximum of 6 cycles of chemotherapy in the absence of tumor progression or unacceptable toxicities.
  Interventions: Drug: Docetaxel; Drug: Sunitinib

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 75mg/m2 day 1, every 3 weeks
Drug: Sunitinib — 7 days of sunitinib 12.5mg orally daily during each cycle
  Arms: Docetaxel + Sunitinib

SUMMARY:
This study aims to find out whether the effect of docetaxel chemotherapy may be improved by combining it with another anti-cancer drug called sunitinib, which stops blood vessels from growing (anti-angiogenic agent). Sunitinib is an oral anti-angiogenic drug that has been approved for the treatment of kidney cancer, a rare form of soft tissue tumor called gastrointestinal stromal tumor, and a rare form of cancer in the pancreas called pancreatic neuroendocrine tumor. Sunitinib is usually given continuously at a dose of 37.5mg (3 pills) daily either alone or in combination with chemotherapy. However, there are studies which have shown that the continuous administration of sunitinib may reduce chemotherapy effectiveness. On the other hand, a short course of sunitinib before each chemotherapy cycle may sensitize the tumor to chemotherapy. This treatment strategy will be used in patients with different kinds of cancers with a commonly used chemotherapy drug, docetaxel. Ths study aims to evaluate if intermittent administration of low dose sunitinib before docetaxel chemotherapy can improve the treatment response in cancer patients.

Study Hypothesis: Low dose, short course sunitinib at 12.5mg daily orally for 1 week prior to chemotherapy can normalize tumor vasculature and enhance delivery of chemotherapy into the tumor, and improve treatment response and progression-free survival.

DETAILED DESCRIPTION:
This is a single-centre, phase II randomized study. Eligible patients will be randomized to docetaxel with or without intermittent sunitinib. A total of eighty patients with measurable tumor will be enrolled over a period of 24-36 months. Eligible patients will be randomized 1:1 to either arm A or arm B. Patients will be stratified according to site of primary tumor (breast vs non-small cell lung cancer vs others) for randomization purposes.

Arm A (Control arm):

Docetaxel 75mg/m2 day 1, every 3 weeks

Arm B (Experimental arm):

Docetaxel 75mg/m2 day 1, every 3 weeks, preceded by 7 days of sunitinib 12.5mg orally daily during each cycle.

Patients will be treated for a maximum of 6 cycles of chemotherapy in the absence of tumor progression or unacceptable toxicities.

Patient will be evaluated weekly for toxicity assessments and full blood count during cycle 1, and on days 1 and 15 of each subsequent cycle.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years.
* Histologic or cytologic diagnosis of carcinoma.
* Measurable tumor, defined as clinically palpable tumor with both diameters 2.0cm or greater as measured by caliper, or radiologically measurable tumor on CT scan with the largest diameter >= 1cm.
* Eastern Cooperative Oncology Group 0-1
* Estimated life expectancy of at least 12 weeks.
* Adequate organ function including the following:

  - Bone marrow: Absolute neutrophil (segmented and bands) count (ANC) >= 1.5 x 109/L Platelets >= 100 x 109/L

  - Hepatic: Bilirubin <= 1.5 x upper limit of normal (ULN), ALT or AST <= 2.5x ULN, (or <=5x with liver metastases)

  - Renal: Creatinine <= 1.5x ULN
* Signed informed consent from patient or legal representative.
* Patients with reproductive potential must use an approved contraceptive method if appropriate (e.g., intrauterine device, birth control pills, or barrier device) during and for three months after the study. Females with childbearing potential must have a negative serum pregnancy test within 7 days prior to study enrollment.

Exclusion Criteria:

* Treatment within the last 28 days with any investigational drug.
* Concurrent administration of any other tumor therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy.
* Major surgery within 28 days of study drug administration.
* Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
* Pregnancy.
* Breast feeding.
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
* Active bleeding disorder or bleeding site.
* Non-healing wound.
* Poorly controlled diabetes mellitus.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* Symptomatic brain metastasis.
* History of significant neurological or mental disorder, including seizures or dementia.
* Known history of systemic connective tissue diseases (e.g., systemic lupus erythematosus, rheumatoid arthritis, systemic sclerosis), vasculities (e.g., giant cell arteritis, Kawasaki disease, Wegener's granulomatosis, Churg-Strauss disease) or sickle cell disease.
* Known history of renal impairment, defined as a Glomerular Filtration Rate (GFR) of less than 30ml/minute.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-05; Primary Completion 2017-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 18 weeks
Clinical benefit rate | 18 weeks
  Clinical benefit rate is defined as the proportion of patients who achieved complete response, partial response, or stable disease for at least 12 weeks, as the best response.

SECONDARY OUTCOMES:
Progression-free survival | 18 weeks until documented disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Soo Chin Lee, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore, Singapore
  - National University Hospital, Singapore

REFERENCES:
- [Background] Bergh J, Bondarenko IM, Lichinitser MR, Liljegren A, Greil R, Voytko NL, Makhson AN, Cortes J, Lortholary A, Bischoff J, Chan A, Delaloge S, Huang X, Kern KA, Giorgetti C. First-line treatment of advanced breast cancer with sunitinib in combination with docetaxel versus docetaxel alone: results of a prospective, randomized phase III study. J Clin Oncol. 2012 Mar 20;30(9):921-9. doi: 10.1200/JCO.2011.35.7376. Epub 2012 Feb 13. PMID 22331954
- [Derived] Ang YLE, Ho GF, Soo RA, Sundar R, Tan SH, Yong WP, Ow SGW, Lim JSJ, Chong WQ, Soe PP, Tai BC, Wang L, Goh BC, Lee SC. A randomized phase II trial evaluating the addition of low dose, short course sunitinib to docetaxel in advanced solid tumours. BMC Cancer. 2020 Nov 17;20(1):1118. doi: 10.1186/s12885-020-07616-4. PMID 33203399